CLINICAL TRIAL: NCT06919328
Title: Absorption and Tolerability of Injectable Administration of Niagen®+, Nicotinamide Riboside Chloride, a Specialized Form of Vitamin B3, as Compared to NAD+: a Double Blinded, Randomized, Controlled Clinical Trial
Brief Title: Absorption and Tolerability of Injectable Administration of Niagen®+, as Compared to NAD+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Collaborators: ChromaDex, Inc. (Industry)
Responsible Party: Principal Investigator, Jessie Hawkins, PhD, Nutraceuticals Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 24-09-1300
Record Dates: First submitted 2025-03-19; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy Aging
Keywords: NAD+
MeSH Terms: interventions — nicotinamide-beta-riboside; NAD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- NR via IM injection (Experimental): 100mg NR 2ml bacteriostatic water via intramuscular (IM) injection
  Interventions: Dietary Supplement: Niagen®
- NR via subcutaneous injection (Experimental): 100mg NR 2ml bacteriostatic water via subcutaneous (SQ) injection
  Interventions: Dietary Supplement: Niagen®
- NR via IV push (Experimental): 100mg NAD+ 2ml bacteriostatic water via intravenous push (IVP) injection
  Interventions: Dietary Supplement: Niagen®
- NAD+ via IM injection (Active Comparator): 100mg NAD+ in 2ml bacteriostatic water via intramuscular (IM) injection
  Interventions: Other: NAD+
- NAD+ via subcutaneous injection (Active Comparator): 100mg NAD+ in 2ml bacteriostatic water via subcutaneous (SQ) injection
  Interventions: Other: NAD+
- NAD+ via IV push (Active Comparator): 100mg NAD+ 2ml bacteriostatic water via intravenous push (IVP) injection
  Interventions: Other: NAD+
- placebo via IM injection (Placebo Comparator): 2ml bacteriostatic water via intramuscular (IM) injection
  Interventions: Other: Placebo
- placebo via subcutaneous injection (Placebo Comparator): 2ml bacteriostatic water via subcutaneous (SQ) injection
  Interventions: Other: Placebo
- placebo via IV push (Placebo Comparator): 2ml bacteriostatic water via intravenous push (IVP) injection
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Niagen® — nicotinamide riboside
  Arms: NR via IM injection; NR via IV push; NR via subcutaneous injection
Other: NAD+ — Nicotinamide adenine dinucleotide
  Arms: NAD+ via IM injection; NAD+ via IV push; NAD+ via subcutaneous injection
Other: Placebo — bacteriostatic water
  Arms: placebo via IM injection; placebo via IV push; placebo via subcutaneous injection

SUMMARY:
This study evaluates the subjective effects of injection administration of NR on healthy adult populations.

DETAILED DESCRIPTION:
The purpose of this work is to explore the tolerability of Niagen®, nicotinamide riboside chloride, a specialized form of vitamin B3, via intramuscular (IM), subcutaneous (SQ), and intravenous-push (IVP) administration, in comparison to NAD+, an active comparator, administered through the same routes.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness and demonstrated ability to comply with all study procedures, as well as availability for the duration of the study
* Lives within 100 miles of the NRI study site
* Any gender, aged 40-65, inclusive
* Good general health as evidenced by medical history
* BMI 25-34.9 kg/m2
* Sedentary behavior (defined as <20 minutes per day or 100 minutes per week of moderate to vigorous exercise)
* Demonstrated fatigue (Fatigue Assessment Scale) defined as a below-average score
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional month after the end of the study
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Current diagnosis of any seizure disorder, diabetes or insulin resistance, any kidney or liver disorder, heart disease, anemia, cancer, or Parkinson's disease
* ANY chronic illness (pre-disease state acceptable)
* Out of range phosphate levels at baseline
* BMI less than 25 or greater than or equal to 35
* Pregnancy, trying to conceive, or breastfeeding
* Known allergic reactions to any components of the intervention or related compounds, including any form of B3
* Positive COVID-19 test within 30 days of the study period
* Recent dramatic weight changes (10% change in body weight in the last 6 months)
* Existing usage of a NAD+ or NAD precursor supplement in any form (oral, nasal, patch, or injection/IV administration), including a B-complex supplement, within 60 days of the study, not including multivitamins.
* Introducing a new medication, supplement, investigational drug, or other intervention (including lifestyle changes) within 60 days of the start of the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
McGill Pain Questionnaire | 1 minute after injection is complete
  The MPQ contains 78 pain related terms to identify the quantity and type of pain experienced. This multi-dimensional tool has three components; sensory, cognitive, emotional. Higher scores indicate higher levels of pain.
Subjective Discomfort | 1 minute after injection is complete
  Subjective discomfort is measured using open-ended questions to qualitatively assess participant comfort during injection.

SECONDARY OUTCOMES:
C-reactive protein | baseline, 90 minutes post injection, day 10
  CRP in serum
Sed Rate | baseline, 90 minutes post injection, day 10
  erythrocyte sedimentation rate through whole blood
plasma viscosity | baseline, 90 minutes post injection, day 10
  Plasma viscosity was measured through blood plasma.

OTHER OUTCOMES:
NRI Sleep Scale | Baseline, Day 10
  The NRI Sleep scale is a validated scale that measures 6 domains of sleep via a Likert scale. Higher scores indicated greater sleep disturbances.
NRI Energy Scale | Baseline, Day 10
  The NRI Energy scale is a validated scale that measures 6 domains of fatigue via a Likert scale. Higher scores indicated greater fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutraceuticals Research Institute, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: No